CLINICAL TRIAL: NCT01180023
Title: Membrane Sweeping in GBS Positive Patients at 37 Weeks Gestation: A Randomized Controlled Trial
Brief Title: Membrane Sweeping in Group B Streptococcus (GBS) Positive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Jennifer Keller, Assistant Professor- OBGYN, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JKeller01
Record Dates: First submitted 2010-05-26; First posted 2010-08-11 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Group B Streptococcus
Keywords: GBS; Membrane sweeping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sweeping (Experimental)
  Interventions: Procedure: Sweeping
- No sweeping (No Intervention)

INTERVENTIONS:
Procedure: Sweeping — Sweeping of membranes during digital exam
  Arms: Sweeping

SUMMARY:
Sweeping or stripping of the membranes (in this paper referred to as "membrane sweeping") is a widely utilized technique to hasten delivery for women at 37+ weeks gestation. The process of membrane sweeping probably causes release of prostaglandins from the decidua and the cervix. The efficacy of membrane sweeping is well studied, and has been shown to increase the number of patients in labor within 72 hours, reduce the frequency of pregnancy continuing beyond 41 or 42 weeks, and reduce the frequency of formal induction of labor. Thus, it is a safe and practical option for women who wish to avoid inductions of labor or postterm pregnancies.

Group B streptococcus (GBS; streptococcus agalactiae) is a gram positive coccus that frequently colonizes the human genital tract. In pregnant women, GBS can cause urinary tract infections, chorioamnionitis, and postpartum endometritis. Newborn infants can also acquire GBS infection during passage through the vagina. Early onset GBS disease in the newborn can lead to pneumonia, meningitis, and sepsis, all of which can be life-threatening. Early onset GBS disease has become rare since the widespread use of GBS screening and prophylactic treatment of pregnant women.

The relationship between early onset GBS disease and sweeping of the membranes is not known. Based on the theoretical increased risk of bacterial seeding after membrane sweeping, as well as concern for fast labors and inadequate treatment after membrane sweeping, some practitioners choose not to sweep membranes in GBS positive patients. A meta-analysis did not show a difference in neonatal or maternal infection rates between women who underwent membrane sweeping and those who did not. ACOG guidelines state "the risks of membrane stripping in GBS positive patients has not been investigated in well-designed, prospective studies. Therefore, data are insufficient to encourage or discourage this practice".

Specific Aims:

In order to help elucidate the effect of membrane sweeping in GBS positive patients, the investigators propose this prospective randomized trial. The investigators primary objective is to determine whether membrane sweeping in GBS positive women is associated with inadequate antibiotic treatment in labor (defined as less than four hours of antibiotic therapy prior to delivery). The investigators secondary objectives are to measure the effect of membrane sweeping on pregnancy duration, length of labor and adverse events potentially related to membrane sweeping such as maternal chorioamnionitis and neonatal morbidity. Randomization is the real research portion of this study, since offering membrane sweeping is already the standard of care. Patients are followed until the time of delivery, which is within 6 weeks of enrollment for most women.

ELIGIBILITY:
Inclusion Criteria:

* All women presenting to the Medical Faculty Associates outpatient Obstetrics clinic who are 37+ weeks
* Are at least 18 years of age and can read and write in English
* Are candidates for vaginal delivery, and qualify for GBS prophylaxis by CDC criteria (any one of the following:

  * have rectovaginal cultures positive for GBS
  * have a GBS UTI this pregnancy
  * have had an infant with GBS disease in a prior delivery) will be offered enrollment in the study.

Exclusion Criteria:

* Patients who are not candidates for vaginal delivery (placenta previa, breech presentation, planned repeat cesarean), will be excluded from the study.
* Patients who are HIV positive will also be excluded, since membrane sweeping may have some risks in these patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Adequate antibiotics received in labor | Data collected from chart after patients delivered, up to 6 weeks after enrollment.
  Charts are reviewed to determine if subjects received appropriate treatment in labor with regards to timing of antibiotic administration

SECONDARY OUTCOMES:
Antibiotics received by neonate | At time of chart review approximately 6 weeks after enrollment
Maternal temperature | At the time of chart review approximately 6 weeks after enrollement
Maternal white blood cell count | At the time of chart reivew approximately 6 weeks after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Keller, MD MPH, Principal Investigator — The George Washington University
Locations (1):
- Medical Faculty Associates, Washington D.C., District of Columbia, United States